CLINICAL TRIAL: NCT07074964
Title: Efficacy of Manual Therapy in Indirect Non-Invasive Neuromodulation of the Vagus Nerve in the Treatment of Bruxism in Young Adult Population up to 40 Years Old
Brief Title: Manual Therapy in Vagus Nerve Neuromodulation for the Treatment of Bruxism
Acronym: TMBruxism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Maider Sánchez Padilla, Principal Investigator, Escoles Universitaries Gimbernat
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMBruxism
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Bruxism, Sleep
Keywords: Sleep Bruxism; Electromyography; Musculoskeletal Manipulations; Vagus Nerve; Autonomic Nervous System; Masticatory Muscles
MeSH Terms: conditions — Sleep Bruxism | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (autonomic nervous system intervention) (Experimental): Manual therapy applied to structures adjacent to the vagus nerve along its pathway (head, neck, thorax, diaphragm, abdomen).
  Interventions: Other: Autonomic nervous system intervention
- Group 2 (control) (Sham Comparator): The hands will be placed on areas similar to those in the intervention group, with the fingertips in contact with the skin of the area. A slight finger pressure will be applied.
  Interventions: Other: Slight finger pressure

INTERVENTIONS:
Other: Autonomic nervous system intervention — Manual therapy applied to structures adjacent to the vagus nerve along its pathway. Head: CV4 tecnique and Jugular foramen tecnique; Neck: stretching and mobilization of the superficial and deep layers; Thorax: Longitudinal and transverse translations of the mediastinum; Diaphragm tecniques, Abdomen: Stretching of the gastro-phrenic ligament with lowering of the stomach and general treatment of the small intestine and the mesentery. Stretching, compression and traction movements will be carried out on these structures.
  Other Names: Intervention
  Arms: Group 1 (autonomic nervous system intervention)
Other: Slight finger pressure — The hands will be placed on areas similar to those in the intervention group, with the fingertips in contact with the skin of the area. A slight finger pressure will be applied, which would not have the same effect as the proposed techniques, since those techniques require a greater intensity of manipulation of the described tissues and structures.
  Other Names: Control
  Arms: Group 2 (control)

SUMMARY:
Introduction:

Sleep bruxism is defined as the repetitive activity of the masticatory muscles, characterized by clenching or grinding of the teeth. Studies confirm the association between sleep bruxism and episodes of masticatory muscle activity, with an increase in autonomic sympathetic activity observed during transient periods of sleep. This is associated with nocturnal awakenings, related to increased cardiac, cerebral (cortical arousal), respiratory, and muscular activity.

Objectives: The main objectives are "To study the mean power frequency (MPF) of the masticatory muscles measured by surface electromyography (sEMG) in the general population (with and without bruxism according to ICSD-3 and DC/TMD criteria)"; and "to assess the effectiveness of manual therapy applied to structures adjacent to the vagus nerve based on its impact on orofacial pain and symptomatology in patients with bruxism".

Material and Methods:

A cross-sectional observational study and a randomized controlled experimental study were designed. The first will analyze data collected by sEMG in the masticatory muscles, at rest and during maximum clenching, comparing results between bruxists and non-bruxists. The second will analyze, compared to the control group, data collected on signs (range of motion alteration, presence of sounds), symptomatology (pain, headaches, sensation of blockage, functional limitation) caused by bruxism, sleep quality (Pittsburgh Sleep Quality Index (PSQI)), oral health-related quality of life (OHIP-14), stress and anxiety status (Perceived Stress Scale and GAD-7 (Generalized Anxiety Disorder-7), respectively), and sympathetic-vagal balance (Heart Rate Variability in its frequency and time domains) before and after a manual therapy intervention on structures adjacent to the vagus nerve pathway (head, neck, thorax, diaphragm, abdomen). The collected data will be analyzed using IBM SPSS® version 25.0.0.

ELIGIBILITY:
Inclusion Criteria:

1. Sleep bruxism diagnosed according to the ICSD-III (International Classification of Sleep Disorders, 3rd edition):

   * Regular or frequent tooth grinding sounds occurring during sleep and the presence of one or more of the following clinical signs and symptoms:

     1. Abnormal tooth wear consistent with reports of clenching/grinding the teeth during sleep
     2. Transient morning pain or fatigue in the jaw muscles; and/or temporal headaches; and/or jaw locking upon awakening, consistent with reports of clenching/grinding the teeth during sleep
2. Sleep bruxism diagnosed according to the RDC/TMD:

   * Interview: During the interview, subjects are asked about the following symptoms: reports of regular or frequent tooth grinding during sleep, muscle fatigue, temporal headache, transient morning muscle pain in the jaw, and jaw locking upon awakening.
   * Physical examination: Presence or signs suggesting abnormal dental wear, such as teeth with flattened cusps and/or loss of contour with dentin exposure.

     * Hypertrophy of the masticatory muscles
     * Dental impressions on the tongue
     * Linea alba on the cheeks along the bite line
     * Damage to dental tissue
     * Excessive dental wear
3. A minimum pain intensity score of 3 on the Visual Analogue Scale at the masseter and temporal algometry points.
4. EMGs with elevated mean power frequency for the masseter and temporalis muscles (to be defined in the first clinical phase-observational study).
5. Age between 18 and 40 years.

Exclusion Criteria:

1. Having suffered direct trauma, mandibular fractures, or surgeries in the orofacial region.
2. Loss of more than 2 teeth, except for the third molar.
3. Use of muscle relaxant medication or medications that may influence motor behavior.
4. Having received botulinum toxin treatment in the last 6 months.
5. Periodontal disorders or current orthodontic treatment or prosthesis.
6. Partial or total dentures.
7. History of medical disorders (severe psychiatric, physiological, or neurological conditions).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Orofacial Pain | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Assessment tests for TemporoMandibular Disorder (TMD) and bruxism condition "AXIS- I" is the assessment tool with a "Symptom questionnaire" that ank about pain in 4 questions.

SECONDARY OUTCOMES:
Orofacial Pain (Masseter and Temporalis) | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with a Pressure Pain Threshold of masseter and temporalis muscles with a DC/ TMD EXAMINATION FORM That measures pain intensity by applying one kilogram of pressure to three points on the temporalis, the masseter, and the temporomandibular joint.
Chronic Orofacial Pain | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Assessment tests for TMD and bruxism condition "AXIS -II" throught the "Graded chronic pain scale version 2.0". It's a self-report questionnaire, typically using a 0-10 numerical rating scale, that evaluates pain intensity and its interference with activities. The GCPS 2.0 classifies patients into different grades of chronic pain from 0 to 4. Higher scores mean a worse outcome.
Range of Motion (subjective) | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Assessment tests for TemporoMandibular Disorder (TMD) and bruxism condition "AXIS- I" is the assessment tool with a "Symptom questionnaire" that ask about mandibular lock.
Range of Motion (Objective) | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Assessment tests for TMD and bruxism condition "AXIS- I" is the assessment tool with aa DC/ TMD EXAMINATION FORM that measures mouth opening, protrusion, and lateral movements in millimeters
Jaw Funcionality | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  "AXIS-II" is the assesment tool that include "Jaw Functional Limitation Scale-20 (JFLS-20)". It consists of 20 items that explore the patient's difficulty in performing various activities related to jaw function. Each item is scored from 0 (no limitation) to 10 (severe limitation). A higher score indicates more functional limitation of the jaw.
Oral behavior | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  "AXIS-II" is the assesment tool that include "The Oral Behavior checklist (OBC)"
Functional impact of Headaches in daily life | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  The assessment will be carried out using HIT-6 (Headeach Impact Test-6). It consists of 6 items that assess key areas affected by headaches. The sum of the responses gives a total score between 36 and 78 points. A higher score indicates more impact and disability due to headache.
Sleep Quality | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Sleep quality is considered one of the most important measures related to bruxism. To assess it, the Pittsburgh Sleep Quality Index (PSQI) questionnaire will be administered. It consists of 19 items answered by the patient and, optionally, 5 additional questions for the bed partner. The 19 items are grouped into 7 components. Each component is scored from 0 (no difficulty) to 3 (severe difficulty). The global score is obtained by summing the 7 components, with a range from 0 to 21 points. A score of 5 or less indicates good sleep quality, while a score above 5 indicates poor sleep quality.
Oral health-related quality of life | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  To assess it, the HIP-14 (Oral Health Impact Profile-14) questionnaire will be administered. It consists of 14 items that explore the frequency of problems related to oral health in daily life. The items are answered on a 5-point Likert scale, ranging from "never" (0 or 1) to "very often" (4 or 5). A higher score indicates worse oral health-related quality of life.
Motor recruitment pattern of the masseter, temporalis, and suprahyoid muscles | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  In resting position and during maximum clenching, as measured by the mean power frequency (MPF) recorded in a surface electromyography.
Stress | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  To assess it, the PSS: Perceived Stress Scale will be administered. It consists of 14 items. It uses a 5-point Likert scale for each item. A higher score indicates more stress.
Anxiety | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  To assess it, the GAD-7 (General Anxiety Disorder-7) will be administered. It consists of 7 items, answered on a 4-point Likert scale. The total score ranges from 0 to 21. A score of 10 or higher is considered the cutoff point for identifying clinically significant anxiety. The higher the score, the greater the anxiety.
Heart Rate Variability (HRV) | From the first assesment (1 week prior to the start of the intervention) to 1 week after the intervention, and data collection on the persistence (1 month, 3 months and 6 months after the end of the intervention). A total of 33 weeks of follow-up.
  Spectral analysis of the time variation between consecutive heartbeats, referred to as the RR interval, which records the activity of the autonomic nervous system. This is collected using the chest strap "Polar H10 Band," which connects to the mobile app "Elite HRV" or "Kubios Software." It collects the frequency measures: LF (low frequency), HF (high frequency), and the ratio between them (LF/HF) as an indicator of sympathetic-vagal balance.
  It collects the time-domain measures: Mean RR interval; SDNN: standard deviation of all RR intervals; pNN50; RMSSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat International de Catalunya (UIC), Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nalamliang N, Sumonsiri P, Thongudomporn U. Masticatory performance is influenced by masticatory muscle activity balance and the cumulative occlusal contact area. Arch Oral Biol. 2021 Jun;126:105113. doi: 10.1016/j.archoralbio.2021.105113. Epub 2021 Mar 30. PMID 33826961
- [Background] Merletti R, Muceli S. Tutorial. Surface EMG detection in space and time: Best practices. J Electromyogr Kinesiol. 2019 Dec;49:102363. doi: 10.1016/j.jelekin.2019.102363. Epub 2019 Oct 19. PMID 31665683
- [Background] Lobbezoo F, Aarab G, Ahlers MO, Baad-Hansen L, Bernhardt O, Castrillon EE, Giannakopoulos NN, Gronbeck A, Hauschild J, Holst-Knudsen M, Skovlund N, Thymi M, Svensson P. Consensus-based clinical guidelines for ambulatory electromyography and contingent electrical stimulation in sleep bruxism. J Oral Rehabil. 2020 Feb;47(2):164-169. doi: 10.1111/joor.12876. Epub 2019 Sep 11. PMID 31430389
- [Background] Lodetti G, Mapelli A, Musto F, Rosati R, Sforza C. EMG spectral characteristics of masticatory muscles and upper trapezius during maximum voluntary teeth clenching. J Electromyogr Kinesiol. 2012 Feb;22(1):103-9. doi: 10.1016/j.jelekin.2011.10.008. Epub 2011 Nov 17. PMID 22100151
- [Background] Berni KC, Dibai-Filho AV, Pires PF, Rodrigues-Bigaton D. Accuracy of the surface electromyography RMS processing for the diagnosis of myogenous temporomandibular disorder. J Electromyogr Kinesiol. 2015 Aug;25(4):596-602. doi: 10.1016/j.jelekin.2015.05.004. Epub 2015 May 27. PMID 26054969
- [Background] Kadioglu MB, Sezer M, Elbasan B. Effects of Manual Therapy and Home Exercise Treatment on Pain, Stress, Sleep, and Life Quality in Patients with Bruxism: A Randomized Clinical Trial. Medicina (Kaunas). 2024 Dec 4;60(12):2007. doi: 10.3390/medicina60122007. PMID 39768887
- [Background] Wojcik M, Siatkowski I. The effect of cranial techniques on the heart rate variability response to psychological stress test in firefighter cadets. Sci Rep. 2023 May 13;13(1):7780. doi: 10.1038/s41598-023-34093-z. PMID 37179419
- [Background] von Piekartz H, Bleiss S, Herzer S, Hall T, Ballenberger N. Does combining oro-facial manual therapy with bruxism neuroscience education affect pain and function in cases of awake bruxism? A pilot study. J Oral Rehabil. 2024 Sep;51(9):1692-1700. doi: 10.1111/joor.13740. Epub 2024 Jun 18. PMID 38894567
- [Background] Matusik PS, Zhong C, Matusik PT, Alomar O, Stein PK. Neuroimaging Studies of the Neural Correlates of Heart Rate Variability: A Systematic Review. J Clin Med. 2023 Jan 28;12(3):1016. doi: 10.3390/jcm12031016. PMID 36769662
- [Background] Perrotta AS, Jeklin AT, Hives BA, Meanwell LE, Warburton DER. Validity of the Elite HRV Smartphone Application for Examining Heart Rate Variability in a Field-Based Setting. J Strength Cond Res. 2017 Aug;31(8):2296-2302. doi: 10.1519/JSC.0000000000001841. PMID 28195974
- [Background] Schaffarczyk M, Rogers B, Reer R, Gronwald T. Validity of the Polar H10 Sensor for Heart Rate Variability Analysis during Resting State and Incremental Exercise in Recreational Men and Women. Sensors (Basel). 2022 Aug 30;22(17):6536. doi: 10.3390/s22176536. PMID 36081005
- [Background] Michalek-Zrabkowska M, Martynowicz H, Wieckiewicz M, Smardz J, Poreba R, Mazur G. Cardiovascular Implications of Sleep Bruxism-A Systematic Review with Narrative Summary and Future Perspectives. J Clin Med. 2021 May 21;10(11):2245. doi: 10.3390/jcm10112245. PMID 34064229
- [Background] Thymi M, Shimada A, Lobbezoo F, Svensson P. Clinical jaw-muscle symptoms in a group of probable sleep bruxers. J Dent. 2019 Jun;85:81-87. doi: 10.1016/j.jdent.2019.05.016. Epub 2019 May 11. PMID 31085350
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Kuang B, Li D, Lobbezoo F, de Vries R, Hilgevoord A, de Vries N, Huynh N, Lavigne G, Aarab G. Associations between sleep bruxism and other sleep-related disorders in adults: a systematic review. Sleep Med. 2022 Jan;89:31-47. doi: 10.1016/j.sleep.2021.11.008. Epub 2021 Nov 19. PMID 34879286
- [Background] Amorim CSM, Espirito Santo AS, Sommer M, Marques AP. Effect of Physical Therapy in Bruxism Treatment: A Systematic Review. J Manipulative Physiol Ther. 2018 Jun;41(5):389-404. doi: 10.1016/j.jmpt.2017.10.014. PMID 30041736
- [Background] Matusz K, Maciejewska-Szaniec Z, Gredes T, Pobudek-Radzikowska M, Glapinski M, Gorna N, Przystanska A. Common therapeutic approaches in sleep and awake bruxism - an overview. Neurol Neurochir Pol. 2022;56(6):455-463. doi: 10.5603/PJNNS.a2022.0073. Epub 2022 Nov 29. PMID 36444852
- [Background] Abe S, Huynh NT, Kato T, Rompre PH, Landry-Schonbeck A, Landry ML, de Grandmont P, Kawano F, Lavigne GJ. Oral appliances reduce masticatory muscle activity-sleep bruxism metrics independently of changes in heart rate variability. Clin Oral Investig. 2022 Sep;26(9):5653-5662. doi: 10.1007/s00784-022-04520-y. Epub 2022 May 10. PMID 35538329